CLINICAL TRIAL: NCT05836662
Title: Comparison of Concussion Education Types
Brief Title: Comparing Concussion Education Types
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Piya Sorcar (Other)
Collaborators: Massachusetts General Hospital (Other); Concordia University Wisconsin (Other)
Responsible Party: Sponsor-Investigator, Piya Sorcar, Founder & CEO, TeachAids
Organization: TeachAids (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2D vs 3D - Concordia
Record Dates: First submitted 2023-04-19; First posted 2023-05-01 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Brain Concussion; Knowledge, Attitudes, Practice
MeSH Terms: conditions — Brain Concussion; Behavior

STUDY DESIGN:
Intervention Model Description: In this randomized study, all participants will receive two types of concussion education (CrashCourse and Brain Fly-Through). Participants will be randomized to the 2D or 3D (Virtual Reality) group, and will experience both concussion educations in that modality (either 2D or 3D).
  During their in person study visit, participants will complete a brief ( ~5 minute) pre-survey before viewing the CrashCourse and Brain Fly-Through concussion educations. Participants will then be asked to complete a brief ( ~2 minute) survey to assess their knowledge, self-efficacy, and empathy surrounding concussions.
  Two months later, participants will receive a brief ( ~5 minute) follow-up survey via email, assessing the same constructs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2D Concussion Education (Active Comparator): During their in person study visit, participants will complete a brief ( ~5 minute) pre-survey before viewing the CrashCourse and Brain Fly-Through concussion educations. Participants in this group will receive both of these educations in 2D (via a video on a laptop). Participants will then be asked to complete a brief ( ~2 minute) survey to assess their knowledge, self-efficacy, and empathy surrounding concussions.
  Interventions: Other: CrashCourse Concussion Education in Virtual Reality
- 3D Concussion Education (Experimental): During their in person study visit, participants will complete a brief ( ~5 minute) pre-survey before viewing the CrashCourse and Brain Fly-Through concussion educations. Participants in this group will receive both of these educations in 3D (via a Virtual Reality headset). Participants will then be asked to complete a brief ( ~2 minute) survey to assess their knowledge, self-efficacy, and empathy surrounding concussions.
  Interventions: Other: CrashCourse Concussion Education in Virtual Reality

INTERVENTIONS:
Other: CrashCourse Concussion Education in Virtual Reality — The TeachAids concussion education, including CrashCourse and Brain Fly-Through, will be shown in 3D (via a Virtual Reality headset). These educations are the exact same content as the 2D versions viewed on a laptop, but the modality (via a VR headset) is different.

SUMMARY:
The purpose of this study is to determine if there are differences in knowledge, self-efficacy, and empathy surrounding concussions, as well as intent to report a concussion, after viewing concussion education (CrashCourse and Brain Fly-Through) in 2D versus in 3D.

In this randomized study, all participants will receive two types of concussion education (CrashCourse and Brain Fly-Through). Participants will be randomized to the 2D or 3D (Virtual Reality) group, and will experience both concussion educations in that modality (either 2D or 3D).

DETAILED DESCRIPTION:
In this randomized study, all participants will receive two types of concussion education (CrashCourse and Brain Fly-Through). Participants will be randomized to the 2D or 3D (Virtual Reality) group, and will experience both concussion educations in that modality (either 2D or 3D).

During their in person study visit, participants will complete a brief ( ~5 minute) pre-survey before viewing the CrashCourse and Brain Fly-Through concussion educations. Participants will then be asked to complete a brief ( ~2 minute) survey to assess their knowledge, self-efficacy, and empathy surrounding concussions.

Two months later, participants will receive a brief ( ~5 minute) follow-up survey via email, assessing the same constructs.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* health professions student (ex: Nursing, PT, OT, Pharmacy, Athletic Training) and/or a student-athlete at Concordia University (Ann Arbor or Mequon campus)

Exclusion Criteria:

- have previously viewed the TeachAids CrashCourse concussion education

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-04-19 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in the participant's knowledge, self-efficacy, and empathy surrounding concussions | 2 months
  Participants will take a pre-survey (prior to receiving the concussion education), an immediate post-survey (right after completion of the concussion education), and two-month post-survey (two months after the concussion education. These surveys will assess participant's knowledge, self-efficacy, and empathy surrounding concussions.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel H Daneshvar, MD, PhD, Principal Investigator — TeachAids and Mass General Brigham
Locations (1):
- Concordia University, Mequon, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No